CLINICAL TRIAL: NCT03309098
Title: Agreement Between Clinician and Instrumented Laxity Assessment
Status: Withdrawn | Type: Observational
Why Stopped: IRB's initial review of this study was not completed and study was withdrawn
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0526-17-EP
Record Dates: First submitted 2017-10-09; First posted 2017-10-13 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Ankle Sprains; Ankle Injuries and Disorders
MeSH Terms: conditions — Ankle Injuries; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ankle Injury: Person who injures their ankle
  Interventions: Diagnostic Test: Ligmaster Arthrometer Assessment

INTERVENTIONS:
Diagnostic Test: Ligmaster Arthrometer Assessment — Perform an anterior drawer, inversion stress test and eversion stress test on the participant with an ankle arthrometer (LigMaster Version 1.26, Sport Tech, Inc, Charlottesville, Virginia).

SUMMARY:
Ankle injuries are the most common acute injury to the active population. It is important to ensure best practices and techniques used in clinics for evaluation are validated and consistent. This study will compare diagnostic outcomes of a clinician and of a diagnostic arthrometer when testing acute ankle injuries.

DETAILED DESCRIPTION:
Ankle injuries, specifically lateral ankle sprains, are the most common acute injury to the active population (Hootman, Dick, & Agel, 2007). It is important to insure the use of best practice and ensure that the techniques being utilized in clinics for evaluation are validated and consistent within the techniques. Manual testing and instrumented testing have not yet been tested within the same cohort.

The purpose of this study is to compare the diagnostic outcomes of a clinician and of a diagnostic arthrometer when testing acute ankle injuries. Participants will be recruited at University of Nebraska at Omahas (UNO) Injury Prevention and Care Clinic and Athletic Training Room in Sapp Fieldhouse. Participants with be members of the UNO Wellness Center or UNO athlete, aged 19-80 years old. During a standard evaluation the participant will have a clinician test manual ligamentous laxity and a blinded clinician testing laxity using an arthrometer. Participation will not alter the normal treatment or care for participants. The author hypothesizes that the diagnostic accuracy for all performed test will be good to excellent when assessed for laxity and moderate to good when assessed for pain.

ELIGIBILITY:
Inclusion Criteria:

* Membership to University of Nebraska at Omahas Wellness Center: a student taking on campus classes or a paying community member. Acute injury occurred within one week of evaluation.

Exclusion Criteria:

* Any condition that is contraindicated for manual test (i.e. fracture).

Ages: 19 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Recreationally active, health adults.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of inversion stress test, eversion stress test and anterior drawer | within 48 hours post-injury
  Assess the diagnostic accuracy of the inversion stress test, eversion stress test and anterior drawer using an arthrometer.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Rosen, PhD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No